CLINICAL TRIAL: NCT05183958
Title: A Multicenter, Randomized Controlled, Phase II Clinical Study of First-line Chemotherapy and Camrelizumab With or Without Radiotherapy in the Treatment of Oligometastatic Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); The First Affiliated Hospital of Wenzhou Medical Univercity (Unknown); Jinhua Municipal Central Hospital (Other); Lishui Municipal Central Hospital (Other Government); The Affiliated People's hospital of Ningbo Univercity (Other); Huizhou Municipal Central Hospital (Other); People's Hospital of Quzhou (Other); Sun Yet-sen Cancer Center (Unknown)
Responsible Party: Principal Investigator, ji yongling, Physician, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2021-389
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined radiotherapy group (Experimental): Chemotherapy :TP program (paclitaxel 175mg/m 2 d1, carboplatin AUC=5 d1 IV Q3W; or paclitaxel 175mg/m 2 d1, cisplatin 75mg/m 2 d1, or paclitaxel 175mg/m 2 d1, cis Platinum 25mg/m 2 d1-3 IV (Q3W, up to 4 cycles). Fluorouracil + cisplatin, cisplatin 80 mg/m 2 d1 IV and 5-Fu 800 mg/m 2 continuous IV d1-5 Q3W (up to 4 cycles).Or cisplatin 50mg/m 2 IV d1; LV 200mg/m 2 IV d1; 5-Fu 2000mg/m 2 24 hours continuous IV d1; or cisplatin 80mg/m 2 IV d1, capecitabine 1000mg/m 2 PO BID d1-14.
  Camrelizumab :200mg every 3 weeks,maximum 6 cycles.
  The experimental group received radiotherapy of the lesion within 8 weeks after the end of chemotherapy and immunotherapy. Immunotherapy shall be started within 8 weeks after the end of all radiotherapy.
  The maintenance immunotherapy of the two groups was: Camrelizumab 200mg Q3W, until PD or toxicity is intolerable or up to 24 months.
  Interventions: Radiation: Radiotherapy group; Drug: Camrelizumab; Drug: Chemotherapy
- Non-radiotherapy group (Placebo Comparator): Chemotherapy :TP program (paclitaxel 175mg/m 2 d1, carboplatin AUC=5 d1 IV Q3W; or paclitaxel 175mg/m 2 d1, cisplatin 75mg/m 2 d1, or paclitaxel 175mg/m 2 d1, cis Platinum 25mg/m 2 d1-3 IV (Q3W, up to 4 cycles). Fluorouracil + cisplatin, cisplatin 80 mg/m 2 d1 IV and 5-Fu 800 mg/m 2 continuous IV d1-5 Q3W (up to 4 cycles).Or cisplatin 50mg/m 2 IV d1; LV 200mg/m 2 IV d1; 5-Fu 2000mg/m 2 24 hours continuous IV d1; or cisplatin 80mg/m 2 IV d1, capecitabine 1000mg/m 2 PO BID d1-14.
  Camrelizumab :200mg every 3 weeks,maximum 6 cycles.
  The control group continued Camrelizumab after 3 weeks of the 4 cycles of chemotherapy combined with immunotherapy.
  The maintenance immunotherapy of the two groups was: Camrelizumab 200mg Q3W, until PD or toxicity is intolerable or up to 24 months.
  Interventions: Drug: Camrelizumab; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiotherapy group — Stereotactic body radiotherapy (SBRT, 8Gy/time, 3 -5 times, if other segmentation schemes are used, recommend BED10 >60Gy) or conventional fractional radiotherapy (parts that are not suitable for SBRT, the total dose is more than 30Gy); the primary lesion should be treated with conventional fractional radiotherapy with a dose of 4000cGy or more;
  Arms: Combined radiotherapy group
Drug: Camrelizumab — 4 cycles for combined therapy. Camrelizumab maintenance.
Drug: Chemotherapy — 4 cycles for combined therapy.

SUMMARY:
A multi-center, open, randomized controlled, phase II clinical study to evaluate the efficiency and safety of chemotherapy and immunotherapy combined with locol radiotharepy in treatment of patients with oligometastatic esophageal carcinoma.

DETAILED DESCRIPTION:
This is a multi-center, open, randomized controlled, phase II clinical study to evaluate the efficiency and safety of chemotherapy and immunotherapy combined with locol radiotharepy in treatment of patients with oligometastatic esophageal carcinoma.For patients required that recurrent or metastatic esophageal cancer, no more than 3 metastatic organs and no more than 5 metastatic lesions. First, all patients receive chemotherapy (the regimen includes paclitaxel and platinum drugs; or cisplatin, pentafluorouracil (5-fluorouracil) ) and other standard first-line chemotherapeutics, combined with Camrelizumab for 4 cycles, and the patients who have not progressed were randomly divided into non-radiotherapy group (control group) and combined radiotherapy group (experimental group) at 1:1 ratio. The experimental group received radiotherapy of the lesion within 8 weeks after the end of chemotherapy and immunotherapy. At least one lesion (both primary and metastatic lesions) was required to be irradiated. Stereotactic body radiotherapy (SBRT, 8Gy/time, 3 -5 times, if other segmentation schemes are used, recommend BED10 >60Gy) or conventional fractional radiotherapy (parts that are not suitable for SBRT, the total dose is more than 30Gy); the primary lesion should be treated with conventional fractional radiotherapy with a dose of 4000cGy or more;The radiotherapy of the primary lesions and metastases focus is carried out at the same time or sequentially, and immunotherapy shall be started within 8 weeks after the end of all radiotherapy. The control group continued Camrelizumab after 3 weeks of the 4 cycles of chemotherapy combined with immunotherapy. The maintenance immunotherapy of the two groups was: Camrelizumab 200mg Q3W, until PD or toxicity is intolerable or up to 24 months. The endpoint are PFS, OS, ORR and toxicity of the two groups .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old, regardless of gender;
2. Histologically or cytologically confirmed recurrent or metastatic esophageal squamous cell carcinoma;
3. Non-regional lymph node metastasis, such as upper neck, retroperitoneal or axillary lymph node metastasis; or distant metastasis, but no more than 3 metastatic organs, and no more than 5 lesions;
4. Patients who have not received other systems of anti-tumor treatment; the patients who have received neoadjuvant/adjuvant and radical concurrent radiochemotherapy, and the last treatment time or progress time exceeds 6 months;
5. Patients who have not progressed after receiving 4 courses of chemotherapy combined with PD-1 immune checkpoint inhibitor treatment (according to the RECIST 1.1 evaluation standard);
6. There are measurable lesions according to the RECIST 1.1 standard (cavity structures such as the esophagus cannot be used as measurable lesions), and the measurable lesions should not have received local treatment such as radiotherapy;
7. ECOG PS score is 0～1;
8. For non-surgically sterilized female patients of childbearing age, the serum or urine HCG test must be negative within 72 hours before randomization;
9. Volunteer to participate in clinical research: fully understand and know the research and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all trial procedures;
10. Have not received immunotherapy or biological therapy before;
11. Hemoglobin ≥90g/L, platelets ≥10×10 9 /L, absolute neutrophil count ≥1.5×10 9 /L;
12. Serum creatinine ≤ 1.5 times UNL;
13. Serum bilirubin≤1.5×UNL, AST (SGOT) and ALT (SGPT)≤2.5×UNL, alkaline phosphatase≤5×UNL;
14. Coagulation function: INR≤1.5 × ULN; if the patient is receiving anticoagulation therapy, PT or APTT is within the acceptable range of treatment;
15. There was no history of interstitial pneumonia or previous interstitial pneumonia.

Exclusion Criteria:

1. In addition to the systemic treatment recommended by this program, patients have received other immune checkpoint inhibitor treatments such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibodies in the past, or any other antibodies or drugs with specific targets for T cell costimulation or checkpoint pathways;
2. Patients have received radiotherapy in the past, and the tumor in the irradiation field has progressed;
3. BMI<18.5kg/m 2 , or weight loss >10% within 2 months before screening ;
4. With brain metastases;
5. With metastasis of the meninges, pleura or pericardium;
6. Esophageal perforation and active esophageal bleeding, with invasion of trachea and large blood vessels in the thoracic cavity;
7. Those who confirmed tumor progression during systemic treatment (RECIST 1.1 standard);
8. Severe symptoms of dysphagia caused by tumor compression require immediate radiotherapy intervention to relieve the obstruction;
9. Systemic treatment toxicity did not return to ≤ CTCAE level 1 (except for hair loss) or the level specified by the inclusion/exclusion criteria;
10. Subjects have cardiovascular diseases or clinical symptoms that are not well controlled, including but not limited to: (1) Heart failure above NYHA II; (2) Unstable angina; (3) Myocardial infarction within 1 year; ( 4) Clinically significant supraventricular tachycardia or ventricular arrhythmia without clinical intervention, or poor control after clinical intervention;
11. Patients with severe lung disease, interstitial pneumonia, or previous history of interstitial pneumonia:
12. Autoimmune diseases (such as: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease), but allow the following diseases to enter the next step of screening: type I diabetes, skin diseases that do not require systemic treatment ( Such as vitiligo, psoriasis);
13. Patients have active hepatitis B (HBV DNA≥2000IU/L or 104copies/ml) or hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of the analysis method);
14. Suffered from an active infection requiring systemic treatment 14 days before the first administration;
15. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection 1 year before enrollment, or patients with active pulmonary tuberculosis infection more than 1 year ago but without formal treatment;
16. Patients with other malignant lesions, except for curable skin cancer (non-melanoma), cervical carcinoma in situ or malignant disease cured ≥ 5 years;
17. Patients who cannot understand the test requirements or may not comply with the test requirements;
18. The investigator believes that some obvious diseases should be excluded from this study;
19. The dose limit of radiotherapy cannot meet the limit requirement set by this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 month
  PFS, defined as the time from randomization to the first occurrence of disease progression.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 month
  The percentage of patients with CR and PR assessed by investigators according to Recist v 1.Subjects evaluated as CR and PR need to be confirmed after 4 weeks (the next curative effect evaluation time specified in the protocol).
Overall survival (OS) | Up to 24 month
  OS, defined as the time from randomization to death due to any cause.
Adverse Events (AEs) | Up to 24 month
  Adverse Events Monitor and evaluate the safety of the treatment during the whole course of treatment and 30 days after the end of the last treatment. If severe toxicity occurs, monitor until 90 days after the end of treatment.According to CTCAE 5.0, the toxicity is classified and recorded.

OTHER OUTCOMES:
Disease Control Rate (DCR) | Up to 24 month
  The proportion of patients who have achieved CR，PR and SD assessed by investigators according to Recist v 1.1.
Duration of Response (DoR) | Up to 24 month
  The duration of overall efficacy refers to the time period from the first evaluation of CR/PR (whichever occurs first) to relapse or PD; the duration of SD refers to the time the subjects were enrolled in this study (The day of enrollment) The time period to PD.

CONTACTS AND LOCATIONS:
Overall Officials: yongling Ji, MD, Principal Investigator — Zhejiang Cancer Hospital; Xianghui Du, MD, Principal Investigator — Zhejiang Cancer Hospital; Ming Chen, MD, Principal Investigator — Sun Yet-sen Cancer Center
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China